CLINICAL TRIAL: NCT00402337
Title: A Randomized, Multicenter, Double-blind, Placebo-controlled, Dose-range-finding, Parallel-group, Phase 2 Trial of Oral Linaclotide Acetate Administered to Patients With Chronic Constipation
Brief Title: Dose-range-finding, Phase 2 Trial of Oral Linaclotide Acetate Administered to Patients With Chronic Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCP-103-201
Record Dates: First submitted 2006-11-18; First posted 2006-11-22 (Estimated); Results first posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-01

CONDITIONS: Chronic Constipation
Keywords: Constipation; Chronic Constipation; Microbia; linaclotide; linaclotide acetate; MD-1100
MeSH Terms: conditions — Constipation | interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 72 ug linaclotide acetate (Active Comparator)
  Interventions: Drug: linaclotide acetate
- 145 ug linaclotide acetate (Active Comparator)
  Interventions: Drug: linaclotide acetate
- 290 ug linaclotide acetate (Active Comparator)
  Interventions: Drug: linaclotide acetate
- 579 ug linaclotide acetate (Active Comparator)
  Interventions: Drug: linaclotide acetate
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: linaclotide acetate — oral, once daily.
  Arms: 145 ug linaclotide acetate; 290 ug linaclotide acetate; 579 ug linaclotide acetate; 72 ug linaclotide acetate
Drug: Matching placebo — oral, once daily
  Arms: Matching Placebo

SUMMARY:
The primary purpose of this study is to evaluate the efficacy and safety of administration of linaclotide acetate in patients with chronic constipation.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Patient meets colonoscopy requirements according to the American Gastroenterological Association
* Patient meets criteria for chronic constipation including weekly bowel movement frequency requirements and reports one or more symptoms of constipation according to protocol requirements
* Patient has successfully completed study requirements with no clinically-significant findings: physical exam, ECG, clinical laboratory tests
* Patient is fluent in English

Exclusion Criteria:

* Patient reports loose or watery stools
* Patient meets criteria for IBS including protocol-defined abdominal discomfort or pain
* Patient may not take prohibited medications per protocol
* Medical diagnoses, medical conditions, or family history that would not make the patient a good candidate for the study or limit the patient's ability to complete the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2006-11; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Microbia Medical Affairs, Study Director — Microbia, Inc.
Locations (58):
- United States (58):
  - Microbia Investigational Site, Huntsville, Alabama
  - Microbia Investigational Site, Tucson, Arizona
  - Microbia Investigational Site, Sherwood, Arkansas
  - Microbia Investigational Site, Anaheim, California
  - Microbia Investigational Site, Sacramento, California
  - Microbia Investigational Site, San Diego, California
  - Microbia Investigational Site, Boulder, Colorado
  - Microbia Investigational Site, Bristol, Connecticut
  - Microbia Investigational Site, Boynton Beach, Florida
  - Microbia Investigational Site, Port Orange, Florida
  - Microbia Investigational Site, Tampa, Florida
  - Microbia Investigational Site, Stockbridge, Georgia
  - Microbia Investigational Site, Peoria, Illinois
  - Microbia Investigational Site, Indianapolis, Indiana
  - Microbia Investigational Site, Clive, Iowa
  - Microbia Investigational Site, Davenport, Iowa
  - Microbia Investigational Site, Louisville, Kentucky
  - Microbia Investigational Site, Monroe, Louisiana
  - Microbia Investigational Site, Silver Spring, Maryland
  - Microbia Investigational Site, Boston, Massachusetts
  - Microbia Investigational Site, Ann Arbor, Michigan
  - Microbia Investigational Site, Traverse City, Michigan
  - Microbia Investigational Site, Olive Branch, Mississippi
  - Microbia Investigational Site, Lincoln, Nebraska
  - Microbia Investigational Site, Great Neck, New York
  - Microbia Investigational Site, Pittsford, New York
  - Microbia Investigational Site, Asheville, North Carolina
  - Microbia Investigational Site, Chapel Hill, North Carolina
  - Microbia Investigational Site, Charlotte, North Carolina
  - Microbia Investigational Site, Fayetteville, North Carolina
  - Microbia Investigational Site, Greensboro, North Carolina
  - Microbia Investigational Site, Raleigh, North Carolina
  - Microbia Investigational Site, Winston-Salem, North Carolina
  - Microbia Investigational Site, Cincinnati, Ohio
  - Microbia Investigational Site, Dayton, Ohio
  - Microbia Investigational Site, Oklahoma City, Oklahoma
  - Microbia Investigational Site, Tulsa, Oklahoma
  - Microbia Investigational Site, Pittsburgh, Pennsylvania
  - Microbia Investigational Site, Sellersville, Pennsylvania
  - Microbia Investigational Site, Anderson, South Carolina
  - Microbia Investigational Site, Columbia, South Carolina
  - Microbia Investigational Site, Simpsonville, South Carolina
  - Microbia Investigational Site, Summerville, South Carolina
  - Microbia Investigational Site, Bristol, Tennessee
  - Microbia Investigational Site, Chattanooga, Tennessee
  - Microbia Investigational Site, Germantown, Tennessee
  - Microbia Investigational Site, Jackson, Tennessee
  - Microbia Investigational Site, Austin, Texas
  - Microbia Investigational Site, Corsicana, Texas
  - Microbia Investigational Site, El Paso, Texas
  - Microbia Investigational Site, San Antonio, Texas
  - Microbia Investigational Site, Ogden, Utah
  - Microbia Investigational Site, Chesapeake, Virginia
  - Microbia Investigational Site, Lynchburg, Virginia
  - Microbia Investigational Site, Olympia, Washington
  - Microbia Investigational Site, Spokane, Washington
  - Microbia Investigational Site, La Crosse, Wisconsin
  - Microbia Investigational Site, Madison, Wisconsin

REFERENCES:
- [Derived] Lembo AJ, Kurtz CB, Macdougall JE, Lavins BJ, Currie MG, Fitch DA, Jeglinski BI, Johnston JM. Efficacy of linaclotide for patients with chronic constipation. Gastroenterology. 2010 Mar;138(3):886-95.e1. doi: 10.1053/j.gastro.2009.12.050. Epub 2010 Jan 4. PMID 20045700

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred over a 13 month period from November 2006 to December 2007 at 57 US study sites.
Pre-assignment Details: Patients went through a 14 to 17 day Pretreatment Period during which the patients provided qualifying bowel habit and symptoms, and rescue medicine usage information through an interactive voice response system (IVRS).
Groups:
- Linaclotide, 72μg: Linaclotide, 72μg dose, oral administration, once per day
- Linaclotide, 145μg: Linaclotide, 145μg dose, oral administration, once per day
- Linaclotide, 290μg: Linaclotide, 290μg dose, oral administration, once per day
- Linaclotide, 579μg: Linaclotide, 579μg dose, oral administration, once per day
- Placebo: Dose-matched placebo, oral administration, once per day.
Period: Overall Study
Arm/Group | Linaclotide, 72μg | Linaclotide, 145μg | Linaclotide, 290μg | Linaclotide, 579μg | Placebo
Started | 59 | 57 | 62 | 63 | 69
Completed | 54 | 51 | 58 | 51 | 61
Not Completed | 5 | 6 | 4 | 12 | 8
Not completed — Adverse Event | 0 | 2 | 2 | 3 | 2
Not completed — Noncompliance | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 5 | 3 | 1 | 6 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0
Not completed — Other Reason | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Linaclotide, 145μg: Linaclotide, 145μg dose, oral administration, once per day. One patient was randomized into the study but did not receive ≥ 1 dose of study drug, thus was not included in the Safety Population.
- Total: Total of all reporting groups
Arm/Group | Linaclotide, 72μg | Linaclotide, 145μg | Linaclotide, 290μg | Linaclotide, 579μg | Placebo | Total
Number analyzed (Participants) | 59 | 56 | 62 | 63 | 69 | 309
Age Continuous [Mean (Standard Deviation); unit: years] | 45.9 (14.1) | 46.4 (11.7) | 48.4 (12.7) | 49.2 (14.0) | 46.1 (15.5) | 47.2 (13.7)
Age, Customized [Number; unit: Participants]
  18 years to 65 years | 52 | 53 | 57 | 57 | 64 | 283
  Older than 65 years | 7 | 3 | 5 | 6 | 5 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 54 | 58 | 56 | 61 | 284
  Male | 4 | 2 | 4 | 7 | 8 | 25
Region of Enrollment [Number; unit: participants]
  United States | 59 | 56 | 62 | 63 | 69 | 309

OUTCOME MEASURES:

1. Primary Outcome: Change From Pretreatment in Weekly Normalized Spontaneous Bowel Movement (SBM) Frequency
Description: Change in SBM frequency during Weeks 1 through 4 of the treatment period from the weekly SBM rate obtained during the pretreatment period.
Time Frame: Change from Baseline to Week 4
Population: 307 patients who received ≥ 1 capsule of study drug and had ≥ 1 post-baseline response to the IVRS Treatment Period Question #12 "How many bowel movements did you have today or yesterday since your last call?" were included in the intent-to-treat (ITT) Population.
Measure: Least Squares Mean (Standard Error); unit: SBMs per week
Arm/Group | Linaclotide, 72μg | Linaclotide, 145μg | Linaclotide, 290μg | Linaclotide, 579μg | Placebo
Number analyzed (Participants) | 59 | 56 | 62 | 62 | 68
SBMs per week | 2.59 (0.407) | 3.25 (0.412) | 3.57 (0.391) | 4.29 (0.394) | 1.45 (0.383)
Statistical Analysis 1: Comparison: Linaclotide, 72μg vs Placebo; The null hypothesis is that the active treatment group is equal to the placebo group; Test type: Superiority or Other; p = 0.0337, ANCOVA
Statistical Analysis 2: Comparison: Linaclotide, 145μg vs Placebo; The null hypothesis is that the active treatment group is equal to the placebo group; Test type: Superiority or Other; p = 0.0010, ANCOVA
Statistical Analysis 3: Comparison: Linaclotide, 290μg vs Placebo; The null hypothesis is that the active treatment group is equal to the placebo group; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 4: Comparison: Linaclotide, 579μg vs Placebo; The null hypothesis is that the active treatment group is equal to the placebo group; Test type: Superiority or Other; p < 0.0001, ANCOVA

2. Secondary Outcome: SBM 75% Responder for the Treatment Period (Based on the Normalized Rate)
Description: A patient was an SBM 75% Responder if the patient was an SBM Responder for ≥3 of the 4 treatment period weeks.
  For each week of the treatment and postreatment periods, a patient was considered an SBM Responder if for that week the patient 1) completed ≥4 days of IVRS questions,2) had an SBM rate of ≥ 3 for the week, and 3) had an increase in SBM rate of ≥ 1 from their baseline weekly SBM rate.
Time Frame: Change from Baseline to Week 4
Population: 307 patients who received ≥ 1 capsule of study drug and had ≥ 1 post-baseline response to the IVRS Treatment Period Question #12 "How many bowel movements did you have today or yesterday since your last call?" were included in the ITT Population.
Measure: Number; unit: participants
Arm/Group | Linaclotide, 72μg | Linaclotide, 145μg | Linaclotide, 290μg | Linaclotide, 579μg | Placebo
Number analyzed (Participants) | 59 | 56 | 62 | 62 | 68
participants | 35 | 31 | 38 | 42 | 22

3. Secondary Outcome: CSBM 75% Responder for the Treatment Period (Based on the Normalized Rate)
Description: A patient was a complete spontaneous bowel movement (CSBM) 75% Responder if the patient was a CSBM Responder for ≥3 of the 4 treatment period weeks.
  For each week of the treatment and postreatment periods, a patient was considered a CSBM Responder if for that week the patient 1) completed ≥4 days of IVRS questions,2) had a CSBM rate of ≥ 3 for the week, and 3) had an increase in CSBM rate of ≥ 1 from their baseline weekly CSBM rate.
Time Frame: Change from Baseline to Week 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Linaclotide, 72μg | Linaclotide, 145μg | Linaclotide, 290μg | Linaclotide, 579μg | Placebo
Number analyzed (Participants) | 59 | 56 | 62 | 62 | 68
participants | 11 | 15 | 20 | 18 | 5

4. Secondary Outcome: Change From Baseline in the Weekly Normalized CSBM Rate for the Treatment Period
Description: CSBMs measured daily during the treatment period. During each daily phone call into the IVRS, patients were asked: How many bowel movements did you have today or yesterday after your last call?
Time Frame: Change from Baseline to Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: CSBMs per week
Arm/Group | Linaclotide, 72μg | Linaclotide, 145μg | Linaclotide, 290μg | Linaclotide, 579μg | Placebo
Number analyzed (Participants) | 59 | 56 | 62 | 62 | 68
CSBMs per week | 1.47 (0.295) | 1.59 (0.298) | 1.75 (0.283) | 2.26 (0.285) | 0.45 (0.279)

5. Secondary Outcome: Change From Baseline in Stool Consistency (BSFS) Score for the Treatment Period
Description: Stool consistency analyses were performed using the 7-point BSFS, whereby a score of 1 = difficult to pass; 2 = sausage shaped but lumpy; 3 = like a sausage but with cracks on surface; 4 = like a sausage or snake, smooth and soft; 5 = soft blobs with clear-cut edges (passed easily); 6 = fluffy pieces with ragged edges, a mushy stool; and 7 = entirely liquid.
Time Frame: Change from Baseline to Week 4
Population: 307 patients who received ≥ 1 capsule of study drug and had ≥ 1 post-baseline response to the IVRS Treatment Period Question #12 "How many bowel movements did you have today or yesterday since your last call?" were included in the ITT. 29 patients with no pretreatment spontaneous bowel movements were excluded from the Stool Consistency analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Linaclotide, 72μg | Linaclotide, 145μg | Linaclotide, 290μg | Linaclotide, 579μg | Placebo
Number analyzed (Participants) | 53 | 53 | 55 | 57 | 60
units on a scale | 1.35 (0.182) | 1.57 (0.177) | 1.68 (0.175) | 2.00 (0.171) | 0.50 (0.170)

6. Secondary Outcome: Change From Baseline in Straining Score for the Treatment Period
Description: Straining was assessed using a 5-point ordinal scale, whereby a score of 1 = not at all, 2 = a little bit, 3 = a moderate amount, 4 = a great deal, and 5 = an extreme amount.
Time Frame: Change from Baseline to Week 4
Population: 307 patients who received ≥ 1 capsule of study drug and had ≥ 1 post-baseline response to the IVRS Treatment Period Question #12 "How many bowel movements did you have today or yesterday since your last call?" were included in the ITT Population. 29 patients with no pretreatment spontaneous bowel movements were excluded from the Straining analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Linaclotide, 72μg | Linaclotide, 145μg | Linaclotide, 290μg | Linaclotide, 579μg | Placebo
Number analyzed (Participants) | 53 | 53 | 55 | 57 | 60
units on a scale | -0.71 (0.102) | -0.97 (0.098) | -1.11 (0.097) | -1.14 (0.095) | -0.52 (0.094)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from November of 2006 to February of 2008.
Arm/Group | Linaclotide, 72μg | Linaclotide, 145μg | Linaclotide, 290μg | Linaclotide, 579μg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/56 | 0/62 | 0/63 | 2/69
Other Adverse Events (participants affected / at risk) | 7/59 | 11/56 | 5/62 | 11/63 | 7/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Linaclotide, 72μg (N=59) | Linaclotide, 145μg (N=56) | Linaclotide, 290μg (N=62) | Linaclotide, 579μg (N=63) | Placebo (N=69)
Humerus fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Linaclotide, 72μg (N=59) | Linaclotide, 145μg (N=56) | Linaclotide, 290μg (N=62) | Linaclotide, 579μg (N=63) | Placebo (N=69)
Abdominal pain (Gastrointestinal disorders) | 2 | 5 | 2 | 2 | 3
Diarrhea (Gastrointestinal disorders) | 3 | 5 | 3 | 9 | 2
Flatulence (Gastrointestinal disorders) | 2 | 3 | 2 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that publication cannot be made for 24 months from the date of final data lock of the study, the sponsor can review the publication prior to public release, sponsor requires a minimum 60 day review period for each publication, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request an additional delay period of 60 days in order to protect potentially patentable information.